CLINICAL TRIAL: NCT05778643
Title: Immunological Mechanisms in the Treatment of Depression and Their Significance in TaKeTiNa Music Therapy as a New Psychotherapeutic Method. A Waitlist-controlled Randomized Group Pilot Study.
Brief Title: TaKeTiNa in the Treatment of Depression: a Pilot Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P066
Record Dates: First submitted 2023-02-21; First posted 2023-03-21 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TaKeTiNa (Experimental): Participants receive TaKeTiNa Music therapy
  Interventions: Behavioral: TaKeTiNa music therapy
- Waiting (No Intervention): Participants receive no additional therapy

INTERVENTIONS:
Behavioral: TaKeTiNa music therapy — TaKeTiNa music therapy uses a group to perform music together. Each member of the group is needed for the synchronization of the whole group. The group actively makes Music with hands, feet, and the voice. At the same time, the therapist frequently introduces new elements into the process and challenges the group in this playful manner. Through this, patients consistently report an increase in mindful awareness and an alleviation of many depressive symptoms, although these effects have not been shown in controlled studies yet.
  Arms: TaKeTiNa

SUMMARY:
The goal of this clinical study's to analyse the impact of TaKeTiNa music therapy in depressed patients.

The main question[s] it aims to answer are:

. Can TaKeTiNa result in a significant pre-to-post intervention decline of depression severity 2. Can TaKeTiNa result in a significantly lower post-intervention depression severity in the T1/T2 group than in the W1/W2 group.

Participants will

* be randomly assigned to the two groups, intervention vs. waitlist
* receive either an eight week TaKeTiNa music therapy or waitlist
* be analysed using questionaires, blood taking, cortisol saliva analysis, measured heart rate variability

Researchers will compare a waitlist to see if TakeTiNa is superior to waitlist

DETAILED DESCRIPTION:
One third of the depressed patients do not respond adequately to conventional treatment. This seems to be associated with increased production of proinflammatory cytokines such as TNF-a and IL-1, as well as dysregulation of cortisol levels. This project aims to investigate Investigate the effectiveness of TaKeTiNa music therapy in the treatment of patients with clinical diagnosis of moderate to severe depression Investigate the physiological and pathophysiological effects of TaKeTiNa using novel blood based biomarkers of depression, especially LDL cholesterol as well as on immune system function in order to establish immune system based biomarkers for better diagnosis and therapy monitoring of major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

Major depressive disorder Ability to walk, speak, and clap

Exclusion Criteria:

* psychotic symptoms
* acute suicidality
* prior intolerance to body therapeutic methods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-14 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of depression severity (HAMD 17) | four month
  Comparison of depression severity (HAMD 17) in the intervention group from beginning of Therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)

SECONDARY OUTCOMES:
Differences in Depression severity (BDI II) | four month
  Differences in Depression severity in the Intervention Group compared to the Control Group , Assessment through BDI II Questionaire
Differences in anxiety (BAI) | four month
  Differences in anxiety in the Intervention Group compared to the Control Group and in comparison to pre-intervention , Assessment through BAI Questionaire
Differences in social anxiety | four month
  Differences in anxiety in the Intervention Group compared to the Control Group and in comparison to pre-intervention , Assessment through social phobia intentory (SPIN), social interaction anxiety scale (SIAS), social phobia scale (SPS)
Differences in enzymes of sphingolipid metabolism | four month
  Differences in enzymes of sphingolipid metabolism in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)
Differences in Composition of adaptive cellular immunity | four month
  Differences in Composition of adaptive cellular immunity in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)
Differences in Adverse events | four month
  Differences in Adverse events in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)
Differences in Mindful Attention and Awareness | four month
  Differences in MAAS in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)
Differences in Resilience | four month
  Differences in RS-25 in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)
Differences in Physical activity | four month
  Differences in Physical activity measured by pedometer in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)
Differences in Heart rate variability | four month
  Differences in Heart rate variability in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)
Differences in Cortisol levels | four month
  Differences in Cortisol levels in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)
Differences in serum lipid levels | four month
  Differences in serum lipid levels in the Intervention Group from beginning of therapy, during the course of therapy, after completion of therapy and after an 8-week follow-up period and in comparison to control group (pre intervention, during intervention, post intervention and after follow up)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia von Zimmermann, MD, Study Chair — UK Erlangen-Nurnberg
Locations (1):
- University Hospital of Erlangen - Psychiatric Clinic, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No